CLINICAL TRIAL: NCT03887091
Title: Use of a Video-based, Personalized Web Page as a Complement to Standard Patient Education for Clinical Trial Participants
Brief Title: Personal Web Page In Clinical Trial Participant Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Mary-Ellen Taplin, MD, Prinicipal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 13-575
Record Dates: First submitted 2019-03-14; First posted 2019-03-22 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Prostate Cancer; Kidney Cancer; Genitourinary Cancer
Keywords: Web Based Tools; Video Communication; Web-based communication
MeSH Terms: conditions — Prostatic Neoplasms; Kidney Neoplasms; Urogenital Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postwire© Virtual Education Cohort (Experimental): * Participants will be administered a brief questionnaire that asks questions about participant internet access, use, and understanding (Appendix B). This questionnaire will be used to determine eligibility.
  * In randomized into the Virtual Education Cohort:A video based, personalized web page will be created that has information related to the participants therapeutic clinical trial.
  * This web page will have videos of a research nurse explaining how to take study medication(s), how to fill out the study drug diary, and a description of the main side effects associated with the study drugs.
  * Clinic Visit Video Recording Cycle 1-4/Day 1
  * Participants from both groups will be asked to complete two surveys before each Day 1 clinic visit for Cycles 1-7
  Interventions: Other: Postwire
- No Video Intervention (No Intervention): Participants will be administered a brief questionnaire that asks questions about participant internet access, use, and understanding (Appendix B). This questionnaire will be used to determine eligibility
  * Participants randomized to the control cohort will follow standard of care procedures involving clinic visits that do not include the use of video or access to a personalized web page.
  * Participants from both groups will be asked to complete two surveys before each Day 1 clinic visit for Cycles 1-7.

INTERVENTIONS:
Other: Postwire — Postwire© is a web-based, video platform
  Arms: Postwire© Virtual Education Cohort

SUMMARY:
This research study is evaluating the effectiveness of video and web-based communication in clinical research compared to standard practices.

DETAILED DESCRIPTION:
Research has shown that many clinical trial participants are confused about clinical trials. Common participant misunderstandings include the idea of randomization, benefits to participants' health, the proven nature of the study intervention, and failure to recognize the primary purpose of the trial. There can sometimes be unintended miscommunication between the study doctor and/or nursing staff and participants. Thus, there is a clear need to identify ways to improve communication during clinical trials. The investigator's current culture of web-based information presentation, whether it takes the form of PowerPoint presentations, videos, websites, or audio tools, suggests that adding such technology to the cancer research realm may improve a participant's clinical trial experience and possibly improve participant understanding and safety while enrolled on a clinical trial. Video and web-based tools in cancer research have the potential to transform clinical trial practice.

ELIGIBILITY:
* Participants must be ≥ 18 years of age
* Participants must have an advanced or metastatic genitourinary malignancy (prostate or kidney cancer)
* Participants must be consented to one of the selected clinical trials (see Appendix A)
* Participants must be able to read and write English
* Participants must have access to the internet at a minimum of once per week
* Participants must use the internet at a minimum of once per week
* Participants must feel at least somewhat confident in how to use the internet, as determined by the eligibility questionnaire to be completed by the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2014-07-21 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Number of cumulative participant caused violations over 4 cycles | 168 Days
  Wilcoxon Rank Sum Test (one-sided alpha = 0.10).

SECONDARY OUTCOMES:
Number of times participants accessed the webpage | 168 Days
  Pearson correlation coefficient (or Spearman, if appropriate
Number of times participants accessed the webpage | 42 Days
  Pearson correlation coefficient (or Spearman, if appropriate
Number of times participants accessed the webpage | 84 Days
  Pearson correlation coefficient (or Spearman, if appropriate
Number of times participants accessed the webpage | 126 Days
  Pearson correlation coefficient (or Spearman, if appropriate)
number of participant-caused protocol violations | 42 Days
  Pearson correlation coefficient (or Spearman, if appropriate)
number of participant-caused protocol violations | 84 Days
  Pearson correlation coefficient (or Spearman, if appropriate)
number of participant-caused protocol violations | 126 Days
  Pearson correlation coefficient (or Spearman, if appropriate)
number of participant-caused protocol violations | 168 Days
  Pearson correlation coefficient (or Spearman, if appropriate)
Participant reported outcomes (PRO) center on treatment satisfaction | PROs collected on Cycle 1 Day 1 and each day 1 of a cycle thereafter until Cycle 7 Day 1, approximately over the course of 7 months.
  FACIT-TS-PS
Participant reported outcomes (PRO) on Perceived Stress | PROs collected on Cycle 1 Day 1 and each day 1 of a cycle thereafter until Cycle 7 Day 1, approximately over the course of 7 months.
  PSS-10

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Ellen Taplin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Requests may be directed to Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu